CLINICAL TRIAL: NCT05577416
Title: A Phase 0/2 Study of AB-218 in Patients With IDH1 Mutated Low Grade Glioma
Brief Title: A Study of AB-218 in Patients With IDH1 Mutated Low Grade Glioma
Acronym: AB-218-IIT-201
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: Walter and Eliza Hall Institute of Medical Research (Other); AnHeart Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022.003
Record Dates: First submitted 2022-09-19; First posted 2022-10-13 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-03

CONDITIONS: Glioma
Keywords: IDH1; Diffuse Astrocytoma; oligodendroglioma; phase 0; perioperative
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma | interventions — Biopsy; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Phase 0 'window of opportunity'/perioperative (Part A) followed by Phase 2 adjuvant treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Safusidenib Erbumine (AB-218) (Experimental): Part A: Peri-operative treatment (Phase 0); Part B: Post operative adjuvant therapy (phase 2)
  Interventions: Procedure: Biopsy; Drug: Part A: Safusidenib Erbumine; Procedure: Surgery (maximal resection); Drug: Part B: Safusidenib Erbumine

INTERVENTIONS:
Procedure: Biopsy — Patients will undergo stereotactic biopsy by craniotomy or burr hole.
Drug: Part A: Safusidenib Erbumine — Part A: Safusidenib Erbumine orally 250 mg BID for 28 days.
Procedure: Surgery (maximal resection) — Surgery: Maximal safe resection, within 24 hours of last dose of Safusidenib Erbumine.
Drug: Part B: Safusidenib Erbumine — Part B: Safusidenib Erbumine orally 250 mg BID for 28 days for a minimum of 12, 28-day cycles subject to ongoing documented evidence of clinical benefit, until disease progression or unacceptable toxicity.

SUMMARY:
The aim of this clinical trial is to evaluate the feasibility of undertaking a Phase 0 surgical study in patients with diagnosis of a IDH1 mutated Low Grade Glioma (LGG) who have not received prior radiation or chemotherapy and are planned to undergo surgical resection.

DETAILED DESCRIPTION:
This is a single arm, open label Phase 0 trial to assess the feasibility, pharmacokinetics and pharmacodynamics of treatment with AB-218 following biopsy and prior to resection in patients with IDH1 mutated glioma.

Participants will receive treatment in 2 parts:

Part A: Biopsy followed by 1 cycle (28 days) of Safusidenib Erbumine (formerly AB-218), an orally available, small molecular inhibitor of mutated IDH1, then safe maximal resection of the tumour.

Part B: Following recovery from surgery, patients will receive at least 12 cycles of Safusidenib, subject to ongoing documented evidence of clinical benefit, until disease progression or unacceptable toxicity.

It is expected that 10 patients will take part in this study.

It is anticipated this research study will enable investigators to objectively measure the biological activity of Safusidenib in patients with IDH1 mutated LGG.

Anti-tumour activity will be assessed by RANO response criteria.

The investigators have previous experience in pre-treating patients with GBM prior to surgery with systemic therapies and collecting tumour, peri-tumour and normal brain tissues for PK, PD and biomarker evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed LGG or new diagnosis of LGG based on MRI
2. Tumours suitable for biopsy and safe for maximal resection in the opinion of the treating neurosurgeon
3. Patients who in the consensus of the treating neurosurgeon require resection of the brain tumour.
4. Patients who do not require immediate definitive resection of the brain tumour in the opinion of the treating neurosurgeon
5. Measurable and/or evaluable disease as per LGG-RANO criteria
6. Age ≥ 18 years of age.
7. ECOG performance score 0-1
8. Life expectancy of at least 24 months, in the opinion of the investigator
9. Adequate haematological, renal and hepatic function
10. Reproductive and contraception criteria as prescribed

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from participation in the study:

1. Patients who require immediate definitive resection due to degree of mass effect or symptoms
2. Multicentric / multifocal tumour
3. Tumour involves cerebellum or brainstem
4. Patients who have undergone surgery for glioma within 24 months of study enrolment
5. Patients who have received prior chemotherapy and / or radiation for a diagnosis of glioma
6. Patients with contraindications to MRI or unwilling to undergo MRI
7. History of central nervous system bleeding as defined by stroke within 6 months before enrolment
8. Evidence of acute intracranial / intra-tumoural haemorrhage, except for participants with stable grade 1 haemorrhage
9. Other general criteria including:

   i) ECG abnormalities ii) significant comorbidity or infection iii) Prior malignancy iv) Recent surgery v) Known allergy or sensitivity to any of the excipients in the investigational product vi) no contraindicated concomitant medications
10. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator would pose a risk to participant safety or interfere with the study evaluation, procedures or completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Phase 0: Feasibility of Phase 0 study in patient population | 14 months
  Number of patients to complete all planned investigations and procedures
Phase 0: pharmacokinetic analysis of tumour tissue | 4 weeks
  Total and unbound AB-218 in tumour tissue
Phase 0: pharmacokinetic analysis of cerebrospinal fluid (CSF) | 4 weeks
  Total and unbound AB-218 in CSF
Phase 2: Number of Adverse events | up to 30 days after last study dose
  Number of adverse events (AEs) according to NCI CTCAE v 5
Phase 2: Incidence of drug related adverse events | up to 30 days after last study dose
  Drug related adverse events
Phase 2: Incidence of dose limiting toxicity | up to 30 days after last study dose
  Dose limiting toxicity events

SECONDARY OUTCOMES:
Phase 0: Incidence of treatment emergent Adverse events | during 1 cycle of AB-128, prior to maximal resection (4 weeks)
  Treatment emergent adverse events (AEs) according to NCI CTCAE v 5
Phase 0: Safety of planned craniotomy and resection after stereotactic biopsy and treatment with AB-218 | 30 days after maximal resection
  30-day morbidity and mortality post surgery
Phase 0: Pharmacodynamic (PD) analysis of AB-218 in tumour | after maximal resection (4 weeks), at progression (optional)
  Changes in 2-hydroxyglutarate (2-HG) levels in tumour
Phase 0: Pharmacodynamic (PD) analysis of AB-218 in cerebrospinal fluid (CSF) | after maximal resection (4 weeks), at progression (optional)
  Changes in 2-hydroxyglutarate (2-HG) levels in cerebrospinal fluid (CSF)
Phase 0: Pharmacodynamic (PD) analysis of AB-218 in plasma | after maximal resection (4 weeks), monthly during treatment, at progression (optional)
  Changes in 2-hydroxyglutarate (2-HG) levels in plasma
Phase 0: anti-tumour activity | 4 weeks
  Objective response (LGG RANO assessment)
Phase 0: Identify factors that can improve the patient experience quality of the service provided to participants using Research Participant Perception Survey short form (RPPS) | 4 months post op
  Understanding the patients' perspective on the peri-operative design and satisfaction with study procedures
Phase 2: Identify factors that can improve the patient experience quality of the service provided to participants using Research Participant Perception Survey short form (RPPS) | 4 months post op
  Understanding the patients' perspective on the peri-operative design and satisfaction with study procedures
Phase 2: anti-tumour activity | 12 weekly until progression
  Objective response (LGG RANO assessment)

OTHER OUTCOMES:
Phase 2: Survival | 30 days after last study dose
  Progression free survival (PFS)
Phase 2: Survival | 30 days after last study dose
  Overall survival (OS)
Phase 2: Survival | 30 days after last study dose
  Time to treatment failure (TTF)
Phase 0: Change in tumour volume in response to Safusidenib | 4 weeks
  Volumetric analysis of post biopsy and pre-op MRI images
Phase 2: Change in tumour volume in response to Safusidenib | 12 weekly until progression
  Volumetric analysis of MRI images during adjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kate Drummond, Prof, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Drummond KJ, Spiteri M, Cain SA, Jones J, Shaya S, Topp M, Lu T, Tobler R, Valkovic AL, Moore Z, Fatunla OE, Kriel J, Moffet JJD, McAlpine H, Rosier M, Guan H, Dimou J, Schadewaldt V, Roberts-Thomson S, McArdle D, Lui E, Voelker-Albert M, di Sanzo S, Nijagal B, Narayana VK, Mitchell CB, Vissers JHA, Grimmond S, Rosenthal MA, Palmer LM, Best SA, Freytag S, Whittle JR. Perioperative IDH inhibition in treatment-naive IDH-mutant glioma: a pilot trial. Nat Med. 2025 Oct;31(10):3451-3463. doi: 10.1038/s41591-025-03884-4. Epub 2025 Aug 21. PMID 40841487
- [Derived] Cain SA, Topp M, Rosenthal M, Tobler R, Freytag S, Best SA, Whittle JR, Drummond KJ. A perioperative study of Safusidenib in patients with IDH1-mutated glioma. Future Oncol. 2024;20(33):2533-2545. doi: 10.1080/14796694.2024.2383064. Epub 2024 Aug 14. PMID 39140289